CLINICAL TRIAL: NCT02719834
Title: An Analgesic Trial to Reduce Pain and Behavior Disruptions in Nursing Home Residents With Alzheimer's Disease
Brief Title: Behavioral Expressions in Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRB201600020; 6AZ10 (Other Grant/Funding Number: Florida Department of Health)
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Last update posted 2018-03-02 (Actual); Status verified 2018-03

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Acetaminophen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acetaminophen, then placebo: Participants in this group will receive acetaminophen for the first four weeks, then placebo for the next four weeks.
  Interventions: Drug: Acetaminophen; Other: Placebo
- Placebo, then acetaminophen: Participants in this group will receive placebo for the first four weeks, then acetaminophen for the next four weeks.
  Interventions: Drug: Acetaminophen; Other: Placebo

INTERVENTIONS:
Drug: Acetaminophen — Acetaminophen (regular strength) will be provided in two capsules: 325 mg, take two capsules 3 times/day for 28 days (1,950 maximum daily dose). Capsules will be labeled to maintain blinding.
  Other Names: Tylenol
Other: Placebo — The placebo will be provided in the same type of capsules as the acetaminophen. Two capsules, given 3x a day for 28 days. Capsules will be labeled to maintain binding.
  Other Names: Methycellulose

SUMMARY:
Behavioral expressions, such as agitation and aggression, affect up to 90% of persons with dementia and are a major source of patient and caregiver distress, nursing home placement, anti-psychotic medication use, restraints, and increased health care costs. The purpose of the research study is to investigate whether reducing pain reduces behavioral expressions of Alzheimer's disease (agitation and aggression).

DETAILED DESCRIPTION:
The research study will investigate if routine analgesic use will reduce behavioral expressions of dementia and pain in older adults with Alzheimer's disease or other dementias. Using a randomized, placebo-controlled, double-blind, cross-over design, the investigators will compare effects of a routine acetaminophen intervention (650 mg administered routinely by mouth three times per day for 4 weeks) to those of routine placebo (methylcellulose), also given for 4 weeks. The maximum dose to be administered will be 1,950 mg per 24 hours, which is below the current FDA recommendations (maximum dose of 3,000 mg/day).

Participants will be randomly assigned to either treatment or placebo group. The initial treatment phase will last for 4 weeks. At the end of the first 4 weeks, the treatment will be reversed after a 3 day washout period. During the 2nd intervention period, the study drug will be reversed (those receiving acetaminophen will receive the placebo drug and vice versa). The second treatment phase will last for 4 weeks. At the end of 2nd treatment phase, all study treatments will be discontinued

ELIGIBILITY:
Inclusion Criteria:

* documented diagnosis of Alzheimer's Disease or other dementia
* history of a typically painful condition, such as osteoarthritis, back pain, or other chronic musculoskeletal pain
* able to swallow oral medication
* history of aggressive or agitated behavior (defined as score of > 39 on the Cohen-Mansfield Agitation Inventory),
* Mini Mental State Exam (MMSE) score < 23

Exclusion Criteria:

* currently taking acetaminophen or opioid medication on a routine (regularly-scheduled, round the clock) basis
* receiving hospice care
* history of liver or renal disease
* drinks more than 3 alcoholic beverages per day
* known allergy or adverse reaction to acetaminophen
* bed-ridden or comatose
* currently taking warfarin

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: We will recruit study participants from senior communities in the Gainesville area.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Mobilization-Observation-Behaviour-Intensity-Dementia Pain Scale (MOBID-2) will be used for changes between the groups at baseline, weeks 2, 4, 6 and 8 | Change from baseline, weeks 2, 4, 6 and 8
  The MOBID-2 is a two-part, observational pain behavior measure. Part 1 assesses pain related to the musculoskeletal system (the most common cause of pain in older adults) during a set of standardized, guided movements during morning care (5 items). Part 2 assesses pain that might originate from internal organs, head, and skin and is monitored over time (5 items). If a pain behavior is detected, pain intensity is rated using a 0-10 numerical rating scale.
Cohen-Mansfield Agitation Inventory (CMAI) will be used for changes between the groups at baseline, weeks 2,4, 6 and 8 | Change from baseline, weeks 2, 4, 6 and 8
  The CMAI is a 29-item instrument designed to measure the frequency with which persons with dementia display agitation and other behavioral disturbances. The measure consists of 4 subscales that measure aggressive behavior (hitting, scratching, cursing), physical non-aggressive behavior (pacing, restlessness, disrobing), verbally agitated behavior (complaining, repetitive questions, negativism) and hiding/hoarding. Item frequency is scored on a 1 to 7 scale, with (1) = never, (2) = < once per week, (3) once or twice per week, (4) several times per week, (5) once or twice per day, (6) several times per day, or (7) several times per hour. Total scores range from 29-203.

CONTACTS AND LOCATIONS:
Overall Officials: Ann Horgas-Marsiske, RN PhD, Principal Investigator — University of Florida
Locations (1):
- Oak Hammock Continuing Care Retirement Faculty, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided